CLINICAL TRIAL: NCT03634787
Title: Heat Shock Proteins: a Pathogenic Driver and Potential Therapeutic Target in Acute Pancreatitis
Acronym: DIAGNON
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Vilnius University (Other)
Responsible Party: Principal Investigator, Aiste Gulla, Senior surgery resident, Vilnius University
Other Study IDs: 158200-17-941-455
Record Dates: First submitted 2018-07-03; First posted 2018-08-16 (Actual); Last update posted 2018-08-16 (Actual); Status verified 2018-08

CONDITIONS: Acute Pancreatitis
Keywords: Heat Shock Proteins, early diagnosis
MeSH Terms: conditions — Pancreatitis; Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and urine samples on admission
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Acute pancreatitis: First time acute pancreatitis. No later than 2 days since the clinical symptoms started.
  Interventions: Diagnostic Test: CT Scan Day 5-7
- Healthy: No major systemic illness

INTERVENTIONS:
Diagnostic Test: CT Scan Day 5-7 — Computed Tomography on Day 5-7 according to a clinical protocol.
  Groups: Acute pancreatitis

SUMMARY:
To investigate the role of Heat Shock Proteins in the mechanism of acute severe pancreatitis. In addition to test the potential treatment target of acute pancreatitis.

All patients who present with clinical symptoms of acute pancreatitis are evaluated for the enrollment of the study.

DETAILED DESCRIPTION:
All patients with acute pancreatitis are evaluated according to modified Atlanta classification acute pancreatitis severity scores.

Blood serum, urine and DNA samples are collected from all patients presented on admission, after 24 hours, 48 hours, 72 hours.

CT is performed in al patients to evaluate necrosis of pancreas Day 5-7 since hospital admission. If necrosis is not present follow-up is stopped.

ELIGIBILITY:
Inclusion Criteria:

* no prior diagnosis of acute pancreatitis
* admission to the hospital within 2 days since the clinical symptoms
* confirmed diagnosis of acute pancreatitis

Exclusion Criteria:

* chronic pancreatitis
* pancreatic cancer

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients admitted to the hospital within 48 hours since the typical symptoms of acute pancreatitis
Sampling Method: Non-Probability Sample
Enrollment: 280 (Estimated)
Dates: Start 2017-10-20 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
To measure the levels of heat shock proteins in serum and plasma in acute severe pancreatitis settings | 2 years
  Different molecular weight Heat Shock proteins role while developing acute pancreatitis.

SECONDARY OUTCOMES:
To measure pancreas cells activity while applying Heat Shock Protein inhibitors | 2 years
  To establish a mechanism explaining the potential use of heat shock proteins inhibitors/ activators for treatment of acute pancreatitis

CONTACTS AND LOCATIONS:
Locations (1):
- Vilnius University Hospital "Santaros Klinikos, Vilnius, Lithuania

IPD SHARING:
Plan to Share IPD: Undecided
We plan to share the data and recruitment status when the study reaches its requirement sample size